CLINICAL TRIAL: NCT04023877
Title: An Open-Label, Single-Dose Study to Determine the Metabolism and Elimination of [14C]E2027 in Healthy Male Subjects
Brief Title: A Study to Determine the Metabolism and Elimination of [14C]E2027 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2027-A001-005
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-07

CONDITIONS: Dementias With Lewy Bodies
Keywords: E2027; [14C]E2027; Dementia with Lewy bodies; Dementia
MeSH Terms: conditions — Lewy Body Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E2027 (Experimental): Participants will receive approximately 130 microcurie (μCi) of [14C]E2027 as a single 50 milligram (mg) (free base), capsule, orally on Day 1.
  Interventions: Drug: E2027

INTERVENTIONS:
Drug: E2027 — E2027 oral capsule.

SUMMARY:
The primary objective of the study is to achieve mass balance recovery of [14C]-radiolabel in urine and feces and to identify and quantify the main elimination pathways of E2027.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

1. Body Mass Index (BMI) of 18 to 30 kilogram per square meter (kg/m^2) at Screening

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from this study:

1. Have participated in a [14C]-research study within the 6 months prior to Day -1
2. Exposure to clinically significant radiation (greater than [>] 100 millisieverts) within 12 months prior to Day -1
3. Clinically significant illness that required medical treatment within 8 weeks or a clinically significant infection that required medical treatment within 4 weeks before dosing
4. Any history of abdominal surgery that may affect pharmacokinetic profiles of study drug (example, hepatectomy, nephrectomy, digestive organ resection but not cholecystectomy nor appendectomy) at Screening or Baseline
5. Any other clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding (including PR > 210 millisecond [msec], QRS > 110 msec), or laboratory test results that required medical treatment at Screening or Baseline
6. A prolonged QT/QTc interval (QTcF > 450 msec) as demonstrated by ECGs at Screening or Baseline
7. Systolic blood pressure > 130 millimetres of mercury (mmHg) or diastolic blood pressure > 85 mmHg at Screening or Baseline
8. Heart rate less than (<) 45 beats per minute (beats/min) or >100 beats/min at Screening or Baseline
9. Known history of clinically significant drug allergy at Screening or Baseline
10. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
11. Known to be human immunodeficiency virus (HIV) positive at Screening
12. Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
13. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug or alcohol test at Screening or Baseline
14. Use of tobacco or nicotine-containing products within 4 weeks before dosing
15. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
16. Engagement in strenuous exercise within 2 weeks before dosing (example, marathon runners, weight lifters)
17. Intake of caffeinated beverages or caffeinated food within 72 hours before dosing
18. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (example, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [example, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard], and charbroiled meats) within 1 week before dosing
19. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing Intake of over-the-counter (OTC) medications within 14 days (or 5 half-lives, whichever is longer) before dosing unless the investigator and sponsor medical monitor consider that they do not compromise participant safety or study assessments
20. Use of any prescription drugs within 4 weeks before dosing
21. Use of illegal recreational drugs
22. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Cumulative Percent of the Radiolabeled Dose of [14C]E2027 in Biological Matrices (Blood, Urine, Feces and Toilet Tissue) | Up to 56 days
  Blood, urine, feces and toilet tissue samples will be collected at specific time points and will be analyzed for the amount of radiolabeled [14C]E2027.
Maximum Concentration (Cmax) of Radiolabeled [14C]E2027, Non-Radiolabeled E2027 and Metabolites in Biological Matrices | Pre-dose up to Day 56 post-dose
Time to Reach Maximum (Peak) Concentration (Tmax) of Radiolabeled [14C]E2027, Non-Radiolabeled E2027 and Metabolites in Biological Matrices | Pre-dose up to Day 56 post-dose
Area Under the Concentration-Time Curve From Time Zero to 24 hours (AUC(0-24h)) of Radiolabeled [14C]E2027, Non-Radiolabeled E2027 and Metabolites in Biological Matrices | Pre-dose up to Day 56 post-dose
Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUC(0-t)) of Radiolabeled [14C]E2027, Non-Radiolabeled E2027 and Metabolites in Biological Matrices | Pre-dose up to Day 56 post-dose
Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC(0-inf)) of Radiolabeled [14C]E2027, Non-Radiolabeled E2027 and Metabolites in Biological Matrices | Pre-dose up to Day 56 post-dose
Terminal Elimination Half-life (t1/2) of Radiolabeled [14C]E2027, Non-Radiolabeled E2027 and Metabolites in Biological Matrices | Pre-dose up to Day 56 post-dose
Apparent Total Body Clearance (CL/F) of E2027 in Biological Matrices | Pre-dose up to Day 56 post-dose
Apparent Volume of Distribution (Vd/F) of E2027 in Biological Matrices | Pre-dose up to Day 28 post-dose
Percent of AUC(0-inf) of Metabolite to E2027 in Biological Matrices | Pre-dose up to Day 28 post-dose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 56 days post-dose
Number of Participants With Clinically Significant Abnormal Laboratory Values | Up to 56 days post-dose
Number of Participants With Clinically Significant Abnormal Vital Sign Values | Up to 56 days post-dose
Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Findings | Up to 56 days post-dose
Number of Participants With Clinically Significant Abnormal Physical Examination Findings | Baseline, Up to 56 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.